CLINICAL TRIAL: NCT01305122
Title: Tumor and Treatments Impact on Neurocognitive Functions and Quality of Life of Patients With OMS Grade II Glioma: Multicentric Prospective Study
Brief Title: Tumor and Treatments Impact on Neurocognitive Functions and Quality of Life of Patients With OMS Grade II Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment too low
Sponsor: Centre Leon Berard (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUMEURS GLIALES
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: OMS Grade II Glioma
Keywords: Glioma; Neurocognitive functions
MeSH Terms: conditions — Glioma | interventions — Mental Status and Dementia Tests; Tea; Stroop Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OMS grade II glioma (Other): neurocognitive tests
  Interventions: Behavioral: neurocognitive tests

INTERVENTIONS:
Behavioral: neurocognitive tests — * inclusion
  * 1 year
  * 3 years
  * 5 years
  Other Names: -MoCA test; - fNART; - Hopkins Verbal Learning test; - Test 10/36; - TEA; - Stroop; - DO80; - VOSP; - Beery; - BDAE; - Token test; - BDI; - STAI; - QLQ-C30 and BN20

SUMMARY:
This is a multicenter prospective study:2 independant cohorts of patients with OMS grade II glioma will be followed during 5 years.

* cohort A: patients in first-line treatment (surgery, radiotherapy or chemotherapy)
* cohort B: patients with disease simple monitoring.

The primary endpoint is to evaluate the impact of tumor and treatments on neurocognitive functions and quality of life, using validate and standard tests.

ELIGIBILITY:
Inclusion Criteria:

* OMS grade II glioma
* signed informed consent
* age >=18
* IK >=80%
* ability to read, write and undertand French

Exclusion Criteria:

* glioma localized to brainstem
* other neurologic or psychiatric disease
* history of other malignancies, other than curatively treated in-situ carcinoma of the cervix or basal cell carcinoma of the skin, or any other curatively treated cancer with no sign of recurrence within 5 years prior to randomization
* neuroleptic concomitant treatment
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-02; Primary Completion 2018-10-21 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
MoCA test | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre SUNYACH, MD, Principal Investigator — Centre Léon Bérard, Lyon - FRANCE
Locations (21):
- France (21):
  - CH Amiens-Picardie, Amiens
  - Institut de Cancérologie de l'Ouest, Angers
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Saint André, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHRU de Lille, Lille
  - Hôpital d'instruction des armées Desgenettes, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital Guy de Chauliac, Montpellier
  - Hôpital Central de Nancy, Nancy
  - Hôpital Pasteur, Nice
  - Centre Antoine Lacassagne, Nice
  - Hôpital Pitié Salpêtrière, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Maison Blanche, Reims
  - CHU Charles NICOLLE, Rouen
  - Centre Henri Becquerel, Rouen
  - Centre René Gauducheau, Saint-Herblain
  - CH Valenciennes, Valenciennes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy